CLINICAL TRIAL: NCT04440878
Title: The Acute Effects of Different Hamstring Muscle Stretching Techniques on Reducing Muscle Resistance to Movement by Ultrasound Elastography
Brief Title: The Acute Effects of Different Stretching Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuksek Ihtisas University (Other)
Responsible Party: Principal Investigator, Kamile UZUN AKKAYA, Principal Investigator, Yuksek Ihtisas University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Kamile UZUN AKKAYA
Record Dates: First submitted 2020-06-17; First posted 2020-06-22 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Muscle Stretching Exercises; Hamstring Muscles
Keywords: Hamstrings; Stretching exercises; Ultrasound elastography
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Static stretching (Experimental): Static stretching will be administered to the hamstring muscles in the first group.
  Interventions: Behavioral: Static stretching
- Mulligan TSLR technique (Experimental): The Mulligan TSLR technique will be administered on the same muscle in the second group.
  Interventions: Behavioral: Mulligan TSLR technique

INTERVENTIONS:
Behavioral: Static stretching — Static stretching exercise will be performed under the supervision of a physiotherapist as 30 seconds of stretching and 15 seconds of rest with 10 repetitions, and the individuals will be asked to participate in the exercise actively.
  Arms: Static stretching
Behavioral: Mulligan TSLR technique — Mulligan TSLR will be applied by a physiotherapist in 3 repetitions with the patient in the supine position.
  Arms: Mulligan TSLR technique

SUMMARY:
The flexibility of the hamstring muscles is very important and many stretching methods are applied on the hamstring muscles for reducing muscle resistance on movement. The objective of this study was to investigate the acute effects of static stretching and the Mulligan traction straight leg raise (TSLR) technique administered to the hamstring muscles on reducing its resistance to movement by using ultrasound elastography in healthy individuals.

DETAILED DESCRIPTION:
The study will be included 22 healthy male volunteers. Static stretching will be administered to the hamstring muscles in the first group and the Mulligan TSLR technique will be administered on the same muscle in the second group. Active knee extension angles of the individuals will be evaluated by a digital goniometer and muscle elasticity will be assessed by ultrasound elastography.

Acute effects of Mulligan TSLR on reducing muscle resistance to movement will be evaluated by ultrasound elastography for the first time in this study. In our study, it was planned to examine the acute effects of static stretching and Mulligan TSLR techniques on reducing muscle resistance to movement by ultrasound elastography in healthy individuals with hamstring shortness.

ELIGIBILITY:
Inclusion Criteria:

* Participants with short hamstring muscles (active knee extension angle below 70 degree),
* Without knee, hip, ankle, or waist pathology,
* Who had not undergone any surgery on the lower extremity were included in the study.

Exclusion Criteria:

* Individuals with musculoskeletal, neurological, or vestibular problems,
* Bone pathologies,
* Joint laxity,
* Diabetes,
* Metabolic syndrome,
* Arthritic or inflammatory problems were excluded.

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-05 (Actual)

PRIMARY OUTCOMES:
The evaluation of muscle flexibility | Five minutes after the application
  The evaluation of muscle flexibility will be made using the ultrasound elastography method by a radiologist.

SECONDARY OUTCOMES:
Range of motion (ROM) | Five minutes after the application
  Active knee extension angles of the individuals will be measured using a digital goniometer by a physiotherapist.

CONTACTS AND LOCATIONS:
Locations (1):
- Yuksek Ihtisas University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cini A, de Vasconcelos GS, Lima CS. Acute effect of different time periods of passive static stretching on the hamstring flexibility. J Back Musculoskelet Rehabil. 2017;30(2):241-246. doi: 10.3233/BMR-160740. PMID 27472859
- [Background] Kerkhoffs GM, van Es N, Wieldraaijer T, Sierevelt IN, Ekstrand J, van Dijk CN. Diagnosis and prognosis of acute hamstring injuries in athletes. Knee Surg Sports Traumatol Arthrosc. 2013 Feb;21(2):500-9. doi: 10.1007/s00167-012-2055-x. Epub 2012 May 24. PMID 22622781
- [Background] Rancour J, Holmes CF, Cipriani DJ. The effects of intermittent stretching following a 4-week static stretching protocol: a randomized trial. J Strength Cond Res. 2009 Nov;23(8):2217-22. doi: 10.1519/JSC.0b013e3181b869c7. PMID 19826305
- [Background] Yildirim MS, Ozyurek S, Tosun O, Uzer S, Gelecek N. Comparison of effects of static, proprioceptive neuromuscular facilitation and Mulligan stretching on hip flexion range of motion: a randomized controlled trial. Biol Sport. 2016 Mar;33(1):89-94. doi: 10.5604/20831862.1194126. Epub 2016 Feb 8. PMID 26929476
- [Background] Umegaki H, Ikezoe T, Nakamura M, Nishishita S, Kobayashi T, Fujita K, Tanaka H, Ichihashi N. Acute effects of static stretching on the hamstrings using shear elastic modulus determined by ultrasound shear wave elastography: Differences in flexibility between hamstring muscle components. Man Ther. 2015 Aug;20(4):610-3. doi: 10.1016/j.math.2015.02.006. Epub 2015 Mar 2. PMID 25795108